CLINICAL TRIAL: NCT01385124
Title: Safety and Efficacy of Oral Cannabidiol for GVHD Prophylaxis in Allogeneic Stem Cell Transplantation
Brief Title: Cannabidiol for Graft Versus Host Disease (GVHD) Prophylaxis in Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6276
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2012-09

CONDITIONS: Graft Versus Host Disease
Keywords: Cannabidiol; GVHD; Allogeneic transplantation; Prophylaxis
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Cannabidiol (Experimental): Oral Cannabidiol 10 mg twice daily will be given from conditioning starting day and until day +30 after allogeneic transplantation. Dose can be doubled every 7 days if no significant side effects documented.
  Interventions: Drug: Oral Cannabidiol

INTERVENTIONS:
Drug: Oral Cannabidiol — Cannabidiol will be dissolved in oil to a predefined concentration. Patients will be given oral cannabidiol 10 mg twice daily from conditioning starting day and until day +30 after allogeneic transplantation.

SUMMARY:
Graft versus host disease (GVHD) is one of the major causes of death in patients undergoing allogeneic hematopoietic cell transplantation. Despite prophylactic measures, the incidence of acute GVHD is estimated at 40-60% among patients receiving transplant from HLA-identical sibling donors, and may even reach 75% in patients receiving HLA-matched unrelated transplants. More effective prevention and treatment strategies are needed.

The immunomodulatory and anti-inflammatory properties of Cannabinoids have been shown in animal models of various inflammatory diseases including multiple sclerosis, inflammatory bowel disease and rheumatoid arthritis.

Cannabidiol is a major non-psychoactive cannabinoid, which has potent anti-inflammatory and immunosuppressive effects.

As such, it may reduce the incidence and severity of GVHD after allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing allogeneic stem cell transplantation.
2. No previous history of psychosis. -

Exclusion Criteria:

1. Previous history of psychosis.
2. Consumption of cannabis during the last 2 moths before transplantation. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall percentage of patients with acute GVHD at day 100 post-transplant | day 100

SECONDARY OUTCOMES:
Percentage of patients with grade III/IV acute GVHD at day 100 post-transplant | day 100

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Yeshurun, MD, Principal Investigator — Davidoff cancer center, Beilinson hospital, Rabin Medical Center
Locations (1):
- Davidoff Cancer Center, Beilin hospital, Rabin medical center, Petah Tikva, Israel

REFERENCES:
- [Derived] Yeshurun M, Shpilberg O, Herscovici C, Shargian L, Dreyer J, Peck A, Israeli M, Levy-Assaraf M, Gruenewald T, Mechoulam R, Raanani P, Ram R. Cannabidiol for the Prevention of Graft-versus-Host-Disease after Allogeneic Hematopoietic Cell Transplantation: Results of a Phase II Study. Biol Blood Marrow Transplant. 2015 Oct;21(10):1770-5. doi: 10.1016/j.bbmt.2015.05.018. Epub 2015 May 30. PMID 26033282